CLINICAL TRIAL: NCT05009927
Title: Randomized, Multicentre, Phase II Study Evaluating the Interest of Imatinib Treatment Maintenance or Interruption After at Least 10 Years of Treatment in Patients With Locally Advanced/Metastatic Gastrointestinal Stromal Tumors (GISTs)
Brief Title: Efficiency of Imatinib Treatment After 10 Years of Treatment in Patients With Gastrointestinal Stromal Tumours (GIST) (Gist-Ten)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIST-TEN
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Gastrointestinal Stromal Tumor (GIST); C-KIT Mutation; Advanced Gastrointestinal Stromal Tumor (GIST)
Keywords: Gastrointestinal Stromal Tumors (GIST); Tyrosine kinase inhibitor; Maintenance therapy; Bayesian design; KIT +; Imatinib; Randomisation study
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imatinib interruption (Experimental): Immediate interruption of imatinib until progressive disease. In case of 1st relapse, imatinib will be reintroduced at 400mg/d and further increased at 800mg/d in case of 2nd relapse after re-introduction.
  Interventions: Drug: Imatinib tablets
- Imatinib maintenancce (No Intervention): Maintenance of imatinib at the last dose routinely taken by the patient in the 10-year period prior to randomization (either 300 or 400 mg once daily). In case of progressive disease imatinib will be increased up to 800mg/day.

INTERVENTIONS:
Drug: Imatinib tablets — Imatinib interruption
  Other Names: Glivec
  Arms: Imatinib interruption

SUMMARY:
This is a 2 arms study concerning patients under imatinib treatment for at least 10 years of treatment with locally advanced/metastatic GIST.

In the first arm, patients will discontinue Imatinib treatment. This arm will allow to determine if the re-introduction of Imatinib at relapse is still an efficient treatment for the control of disease.

In the second arm, patients will continue Imatinib treatment, allowing to determine if the continuation of this treatment is efficient for disease control, by the rate of non-progression disease.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors (GISTs) arise from mesenchymal stem cells which also give rise to the interstitial cells of Cajal within the GI tract. A large majority of GIST tumors harbour activating mutations in the proto-oncogenes KIT and/or PDGFRA, both coding cell-surface cytokine receptors with tyrosine-protein kinase activity.

Imatinib mesilate (Glivec®, Novartis Pharma SAS) is a selective tyrosine kinase inhibitor, leading to inhibition of KIT and PDGFRA signalling pathways. The introduction of imatinib has revolutionised the therapeutic management of GIST patients and has provided an unprecedented demonstration of the clinical benefit of a targeted therapy for patients with advanced/metastatic solid tumors.

Several studies have investigated the optimal duration of imatinib treatment in the advanced phase. The BFR14 trial demonstrated that 31% of advanced GIST patients treated with continuous imatinib beyond 1 year had documented disease progression compared to 81% in the interrupted imatinib group (p<0.0001). The authors concluded that treatment interruption resulted in rapid progression in most patients with advanced GIST and therefore should not be recommended in standard practice unless the patient experienced significant toxicity or disease progression. An update of the BFR14 trial at a median follow-up of 37 months showed that 91% of patients in the interrupted arm versus 62% in the continuous arm experienced progressive disease (p<0.0001). Majority (92%) of patients in the interrupted arm achieved tumor control once they recommenced imatinib after first progression. Ray-Coquard et al. reported that stopping imatinib after 5 years resulted in a higher rate of disease progression than imatinib maintenance in patients with advanced GIST responding to or stabilised by imatinib.

However, whether lifelong imatinib treatment duration is mandatory in metastatic GIST patients remains unclear. It is not known whether a cytostatic treatment of 10 years or longer is sufficient to inhibit definitively GIST cancer cells proliferation even after the interruption of the kinase inhibitor. This question has broad implications for all targeted therapies.

The aim of the present study is to address this question rigorously in a randomized setting. The investigators therefore want to determine whether prolonged use of imatinib beyond 10 years is needed to reduce the risk of GIST recurrence and to improve overall survival. For patients with imatinib interruption after at least 10 years of treatment, the investigators want to determine if imatinib rechallenge is efficient for treating recurrence. Therefore, the investigators design an open-label, randomized, multicenter phase II study to determine the clinical impact of maintaining imatinib treatment beyond 10 years in patients with locally advanced/metastatic GIST.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age;
* Histologically documented diagnosis of malignant advanced/metastatic GIST with immunohistochemical documentation of c-kit (CD117) expression either by the primary tumor or metastases;
* Eastern Cooperative Oncology Group (ECOG) - Performance status (PS) 0 to 2 evaluated within 7 days prior to the date of inclusion.
* Patient must be under imatinib treatment (at 300 or 400mg/day) maintained for 10 years or over with no more than 12 months in total or 3 consecutive months of interruption during the treatment period;
* Patient with controlled disease (without any progression under imatinib);
* Willingness and ability to comply with scheduled visits, treatment plans , laboratory tests, and other study procedures;
* Covered by a medical/health insurance;
* Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment.

Exclusion Criteria:

* Patient concurrently using other approved or investigational antineoplastic agents;
* Patient with GIST harboring the mutation D842V in PDGFRA;
* Major concurrent disease affecting cardiovascular system, liver, kidneys, haematopoietic system or else considered as clinically important by the investigator and that could be incompatible with patient's participation in this trial or would likely interfere with study procedures or results;
* Prior history of other malignancies other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of the disease for at least 3 years;
* Patient receiving concurrent treatment with warfarin (acceptable alternative: low-molecular weight heparin) or any prohibited concomitant and/or concurrent medications
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection;
* Major surgery within 2 weeks prior to study entry.
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Pregnant or breastfeeding woman
* Patient requiring tutorship or curatorship or patient deprivied of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free-rate at 6 months (PFR 6m) | 6 months after randomization
  Defined as the rate of patients with a non-progressive disease 6 months after randomization

SECONDARY OUTCOMES:
Progression-free-survival (PFS) | 5 years (i.e. at the the time of last patient last visit)
  Time from the date of randomization to the date of the first documented progression, or date of death due to any cause. Patients with no event at the time of the analysis will be censored at the date of last available tumor assessment
Overall Survival (OS) | 5 years (i.e. at the the time of last patient last visit)
  the time from the date of randomization to the date of death due to any cause.
Safety profile | 5 years (i.e. at the the time of last patient last visit)
  The assessment of safety will be based mainly on the frequency of AE based on the Common Toxicity Criteria version 5
Quality of Life (QoL) | 5 years (i.e. at the the time of last patient last visit)
  QoL will be assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of life Questionnaire (QLQ-C30).
Progression-free survival rechallenge | 5 years (i.e. at the the time of last patient last visit)
  the time from the date of imatinib reintroduction in the experimental arm to the date of subsequent progression, or date of death due to any cause. Patients with no event at the time of the analysis will be censored at the the date of last available tumor assessment.
Objective Response Rate (ORR) after imatinib reintroduction | 5 years (i.e. at the the time of last patient last visit)
  Defined as the proportion of patients with a best overall response of Partial Response (PR) or Complete Response (CR) after imatinib reintroduction
Duration of response (DOR) | 5 years (i.e. at the the time of last patient last visit)
  the time from the date of first objective response following the reintroduction of imatinib to the date of the first subsequent documented radiological progression or death and censored at the date of last available tumor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, Pr, Principal Investigator — Centre Léon Bérard, Lyon
Locations (13):
- France (13):
  - CHU Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - CHU de Reims, Reims
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest - Site Réné Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien NEUWIRTH, Saint-Paul-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Goustave Roussy, Villejuif